CLINICAL TRIAL: NCT04941859
Title: The Study of Chinese Medicine Acuity Patching Combined Massage in the Treatment of Patients With Acute Poisoning and Stomach Washing
Brief Title: Medicine Acuity Patching Combined Massage in the Treatment of Patients With Acute Poisoning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0023
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Poisoning Patients
Keywords: Acute oral intoxication; Acupoint application; Point massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients in the experimental group were treated with acupoint application combined with acupoint massage on the basis of standard treatment for acute poisoning. When the patient began to launder the stomach, the acupoint was applied to Shenque (umbilical). After the end of the gastric launder, Shenque acupoint and Zusanli diarrhea method (referring to counterclockwise and strong stimulation) were massaged for 15 minutes, and the massage frequency was Q8H.
  Interventions: Behavioral: acupoint massage and application
- control group (No Intervention): The treatment plan of control group was carried out according to the diagnosis and treatment standard of acute poisoning.

INTERVENTIONS:
Behavioral: acupoint massage and application — Patients in the experimental group were treated with acupoint application combined with acupoint massage on the basis of standard treatment for acute poisoning. When the patient began to launder the stomach, the acupoint was applied to Shenque (umbilical). After the end of the gastric launder, Shenque acupoint and Zusanli diarrhea method (referring to counterclockwise and strong stimulation) were massaged for 15 minutes, and the massage frequency was Q8H.
  Arms: experimental group

SUMMARY:
This topic in western medicine combined on the basis of gastric lavage therapy in patients with acute poisoning acupoint sticking of traditional Chinese medicine and acupuncture point massage treatment, aims to smoothly accelerate cleaning and discharge poison, increase the poisoning patients rescue success rate, improve patient quality of life, for the clinical treatment of acute poisoning provides a new method of TCM nursing, to further exert TCM nursing characteristics.

DETAILED DESCRIPTION:
With the rapid development of national economy, people's exposure to a variety of chemicals, drugs and other opportunities to increase, the types of substances causing poisoning tend to be diversified, acute poisoning frequently occur. Data showed that in some regions of China, poisoning cases accounted for 2.7%~ 3.6% of the patients admitted to the emergency department in the same period , and 8.3 % of the patients rescued in the emergency department in the same period , and its fatality rate was higher than the total fatality rate in the emergency department . The incidence of poisoning was 18/100,000 in urban residents and 69.22/100,000 in rural areas, accounting for 10.7% of all deaths. Poisoning incident is an important part of national public health emergency management. According to the statistics of China's Ministry of Health in 2013, poisoning has entered the top five major causes of death in China, and the number of acute poisoning cases has been increasing year by year . The diagnosis and treatment of acute poisoning and the effective and rapid treatment have become an important task for emergency clinical workers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with oral acute poisoning who were first diagnosed in our hospital and completed gastric lavage;
2. The skin of umbilical cord and bilateral Zusanli acupoints had no injury, scar, rash and other skin diseases.
3. The patient or the patient's family member signed the informed consent and expressed their willingness to receive treatment.

Exclusion Criteria:

1. Patients with severe conditions requiring cardiopulmonary resuscitation or with severe trauma or multiple injuries;
2. Patients with heart, brain, liver, kidney and hematopoietic system diseases and other serious primary diseases;
3. Patients with a history of gastrointestinal diseases (such as postoperative cancer, intestinal obstruction, and large intestinal polyps) that affect gastrointestinal emptying;
4. Failing to receive treatment according to regulations or taking poison again during hospitalization and unable to judge the curative effect.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
complications | one year
  Incidence of complications within 24 hours of admission: including nausea, vomiting, and abdominal pain
Time of first bowel movement | through study completion, an average of 1 year
  Time of first bowel movement
patient duration of hospital stay | through study completion, an average of 1 year
  patient duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: minfei yang, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No